CLINICAL TRIAL: NCT03717233
Title: Assistive ExoSkeleton & ExoTendon Platform to Enable Wearable Rehabilitation Robotics
Brief Title: Assistive ExoSkeletons to Enable Wearable Rehabilitation Robotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Results Group LLC (Industry)
Collaborators: Southern Connecticut State University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FB20181
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot Ulcer Associated With Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetic Foot | interventions — Exoskeleton Device

STUDY DESIGN:
Intervention Model Description: Participants will be evaluated as their own controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Arm (Experimental): Participants will be used as their own controls. Participants will be evaluated using exo-skeletons with non-motorized spring elements in parallel to the Achilles tendon. Up to 5 different levels of spring force will be evaluated to evaluate the impact upon plantar pressure and measures of fall risk.
  Interventions: Device: Exoskeleton

INTERVENTIONS:
Device: Exoskeleton — Ankle-foot exoskeleton - device to help reduce load on the bottom of the front of the foot

SUMMARY:
Study will evaluate the use of lower-limb assistive exo-skeletons worn on the ankle and foot. Participants will wear the exo-skeletons and walk in a safe environment. Measurements will be taken to determine how the exo-skeletons affect the pressure on the feet of people with diabetic foot ulcer and how they walk.

DETAILED DESCRIPTION:
Study will evaluate the use of lower-limb assistive exo-skeletons worn on the ankle and foot. Participants will include those with self-described history of Diabetic Foot Ulcer and age-matched healthy volunteers. Participants will wear the exo-skeletons and will be asked to walk 32 feet, and to stand quietly for 30 seconds.

Measurements will be taken to evaluate how the exoskeletons affect how people walk, and will also evaluate the pressure on the bottom of their feet. These measurements will be repeated multiple times to evaluate four different exo-tendon spring rates, and two sets of control shoes.

Exo-skeletons have been shown to reduce the pressure on the bottoms of people's feet and to reduce the effort to walk. This study is necessary to understand the contribution of different levels of exo-skeleton spring force to these effects.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported history of diabetic foot ulcer

Exclusion Criteria:

* Unable to continuously ambulate/walk ≥ 40 feet without an assistive device, such as a cane or walker
* Signs/symptoms of an infected foot lesion/ulcer as determined by a basic foot exam
* Trans-metatarsal foot amputation or more significant amputation.
* Symptomatic for signs/symptoms of cardiovascular disease as determined from interpretation of the 2017 PAR-Q+ (predicated on participant responses of "yes" indicating symptomatic/unstable medical conditions to page 2 and page 3 of the 2017 PAR-Q)
* Participants will be excluded from this study if they demonstrate pre-participation, or chronic, signs/symptoms of hypoglycemia: Confusion, unusual headache, unusual visual disturbances, self-reported mental dullness, shakiness, self-reported weakness, abnormal sweating, undue nervousness/anxiety, and/or tingling of the mouth, toes, and/or fingers or if they answer yes to question 5b and 5c of the 2017 PAR-Q+ .
* Participants will be temporarily excluded from this study if they are symptomatic for acute illness such as cold or fever. If the participant is symptomatic for acute illness such as cold or fever, participation will be reconsidered upon illness resolution.
* If participants answer yes to question 4a of the 2017 PAR-Q+ and if they demonstrate pre-study participation resting blood pressure < 90/60 mmHg and >140/90 mmHg .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Forefoot plantar pressure | 30 minutes
  Measurements of the force and pressure on the bottom of the front of the foot

SECONDARY OUTCOMES:
Measures of fall risk | 30 minutes
  Measurements of postural sway, balance and gait speed to provide an indication of participant's risk of falling while wearing different shoes.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rancho Los Amigos, Los Angeles, California
  - Southern CT State University, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roser MC, Canavan PK, Najafi B, Cooper Watchman M, Vaishnav K, Armstrong DG. Novel In-Shoe Exoskeleton for Offloading of Forefoot Pressure for Individuals With Diabetic Foot Pathology. J Diabetes Sci Technol. 2017 Sep;11(5):874-882. doi: 10.1177/1932296817726349. PMID 28859516